CLINICAL TRIAL: NCT00086229
Title: A Pharmacokinetic Study of Glucosamine and Chondroitin
Brief Title: Absorption and Distribution of Glucosamine and Chondroitin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001938-01 (NIH)
Record Dates: First submitted 2004-06-28; First posted 2004-06-29 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Osteoarthritis
Keywords: Complementary Therapies
MeSH Terms: conditions — Osteoarthritis | interventions — Glucosamine; Chondroitin

INTERVENTIONS:
Drug: Glucosamine
Drug: Chondroitin

SUMMARY:
The purpose of this study is to examine the way the dietary supplements glucosamine and chondroitin are absorbed and distributed throughout the body.

DETAILED DESCRIPTION:
Osteoarthritis is the most common musculoskeletal disease in the world. While predisposing conditions have been identified, the actual cause of osteoarthritis remains unknown. Traditional treatments, most often anti-inflammatory drugs and pain relievers, produce variable results and may cause significant toxicity. The use of complementary and alternative therapies in the treatment of osteoarthritis has become more common, and particular interest has focused on glucosamine and chondroitin treatments. This study will examine the pharmacokinetics of glucosamine and chondroitin.

This study consists of two phases. In Phase I, participants will have two study visits, during which multiple blood samples will be taken to determine levels of glucosamine and chondroitin found naturally in the body. During Phase II, participants will be randomly assigned to receive glucosamine, chondroitin, or a combination of the two for 3 months. Blood samples will be taken at each of the three Phase II study visits to examine the pharmacokinetics of glucosamaine and chondroitin.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk

Exclusion Criteria:

* Allergy to glucosamine, chondroitin, or shellfish
* Liver or kidney disease
* Diabetes mellitus
* Concurrent use of other complementary or alternative therapies

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-04; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G. Jackson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States